CLINICAL TRIAL: NCT01404195
Title: High-protein Nutritional Intervention Based on β-hydroxy-β-methylbutirate, Vitamin D3 and Calcium on Obese and Lean Aged Patients With Hip Fractures and Sarcopenia. The HIPERPROT-GER Study.
Brief Title: Hyperprotein Nutritional Intervention in Elderly Patients With Hip Fracture and Sarcopenia
Acronym: HIPERPROT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Viamed Valvanera, Spain (Other)
Collaborators: University of Navarra (Other)
Responsible Party: Principal Investigator, Vincenzo Malafarina, MD MSc, MD MSc, Hospital Viamed Valvanera, Spain
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HVVV-Log-01; HSJDPAM01SARCOP2011 (Other: Hospital San Juan de Dios); ViamedValvaSarcoHF (Other: Hospital Viamed Valvanera)
Record Dates: First submitted 2011-07-22; First posted 2011-07-27 (Estimated); Last update posted 2016-02-05 (Estimated); Status verified 2016-02

CONDITIONS: Sarcopenia; Hip Fracture
Keywords: Nutritional supplement; CaHMB; Barthel index; Frailty
MeSH Terms: conditions — Sarcopenia; Hip Fractures; Frailty

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ensure Plus Advance, Supplement (Experimental): Participating patients will be dispensed two bottles daily, one at breakfast and one in the evening, seven days a week.
  Interventions: Dietary Supplement: Ensure Plus Advance
- Control (No Intervention): without supplementation

INTERVENTIONS:
Dietary Supplement: Ensure Plus Advance — Participating patients will be dispensed two small bottles daily, one at breakfast and one in the evening, seven days a week
  Arms: Ensure Plus Advance, Supplement

SUMMARY:
1. RATIONALE The unique characteristic of our study lies in the attempt to reverse the functional impairment experienced by sarcopenic patients with hip fracture using nutritional intervention. What makes this study different from prior studies is that it will be conducted in a hospital setting, unlike most prior studies, which were conducted in a community setting. The association between muscle mass and strength, inflammatory indices, and functional impairment versus dependence and fragility will also be measured.
2. HYPOTHESIS The hypothesis of our study is that nutritional intervention enriched in metabolites of essential amino acids (beta-hydroxy-beta-methylbutyrate) is effective for treating sarcopenia in elderly patients with hip fracture and improves functional level.
3. OBJECTIVES Primary objective is to assess functional improvement after nutritional intervention in sarcopenic patients with hip fracture, as measured using Barthel index.

   Secondary objectives will include: 1) to show the relationship between metabolic and inflammatory indices and sarcopenia; 2) to show how sarcopenia and its treatment influence the risk of fall; 3) to show muscle mass improvement; 4) to show increased strength; 5) to assess mortality and morbidity.
4. EXPECTED RESULTS The investigators expect to find that the supplemented group experiences throughout the study period a significant improvement in functional status (Barthel index), an increase in muscle mass, and a reduction in fat mass. An increased strength and a reduction in associated complications (falls) are also expected. The investigators hope to be able to show reductions in inflammatory indices and insulin resistance.

To conclude, by improving muscle strength and mass the investigators expect to find a reduction in the disability and dependence of this population group.

DETAILED DESCRIPTION:
INTRODUCTION Sarcopenia is the loss of muscle mass and function associated to age. Rosemberg first spoke of sarcopenia in 1989. A progressive loss of muscle mass occurs from approximately 40 years of age. This loss is estimated at about 8% by decade until the age of 70 years, after which the loss increases to 15% by decade. Healthcare costs attributable to sarcopenia in the United States (US) in 2000 were estimated to be 18.5 billion dollars.

It would be natural to assume a direct relationship between muscle mass and strength, but loss of muscle mass is not the main mechanism for loss of strength.

Proximal femur (hip) fracture is a substantial cause of morbidity and mortality in the elderly. One-year mortality after a hip fracture ranges from 12% and 37%, with an 11% incidence during the first few months.

Twenty-five percent of elderly patients with hip fracture require institutionalization, at least temporary, and only 40% fully recover their pre-fracture functional status.

Nutritional therapy, particularly beta-hydroxy-beta-methylbutyrate (HMB), a metabolite of the essential amino acid, leucine, has aroused great expectations. All prior studies about nutritional supplementation with HMB have shown an improved muscle metabolism, decreased protein degradation, and a significant increase in fat-free mass in both young and elderly people.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 65 years or older
* Diagnosis of traumatic hip fracture
* Patients admitted for rehabilitation
* Patients signing informed consent.

Exclusion Criteria:

* Stage 4 renal failure
* Child C stage hepatic insufficiency
* Barthel index < 20 in the six months prior to admission
* Dysphagia for liquids
* Active oncological disease who are receiving treatment
* Severe clinical conditions compromising and threatening their lives
* Morbid obesity (BMI > 40)
* BMI < 21 kg/m2
* Albumin levels < 2.1 g/dL
* MNA < 11
* Charlson index ≥ 6
* diabetes mellitus
* Patients not doing rehabilitation.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 110 (Actual)
Dates: Start 2012-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Barthel index | On admission to hospital and at discharge.
  functional improvement after nutritional intervention in sarcopenic patients with hip fracture, as measured using Barthel index.

SECONDARY OUTCOMES:
Change from baseline in bioelectrical impedance analysis | On admission to hospital and at discharge.
  Show muscle mass improvement
Change from baseline in strength will be measured in the dominant hand using a portable JAMAR dynamometer | On admission to hospital and at discharge.
  Show an increased strength
Death for any cause | During admission
  assess mortality and morbidity
Univariate analysis of the relationship between levels of IL-1, IL-6 and TNF-alpha and values of bioelectrical impedance | On admission to hospital and at discharge
  To show the relationship between inflammatory indices and sarcopenia
Prevalence of sarcopenia | hospital admission
  To determine the prevalence of sarcopenia in elderly patients hospitalized for hip fracture.

CONTACTS AND LOCATIONS:
Overall Officials: Vincenzo Malafarina, MD Msc, Principal Investigator — Clinica Los Manzanos, Lardero, Spain; M Angeles Zulet, PhD, Study Chair — University of Navarra
Locations (1):
- Clinica Los Manzanos, Logroño, La Rioja, Spain

REFERENCES:
- [Background] Janssen I, Heymsfield SB, Wang ZM, Ross R. Skeletal muscle mass and distribution in 468 men and women aged 18-88 yr. J Appl Physiol (1985). 2000 Jul;89(1):81-8. doi: 10.1152/jappl.2000.89.1.81. PMID 10904038
- [Background] Cruz-Jentoft AJ, Baeyens JP, Bauer JM, Boirie Y, Cederholm T, Landi F, Martin FC, Michel JP, Rolland Y, Schneider SM, Topinkova E, Vandewoude M, Zamboni M; European Working Group on Sarcopenia in Older People. Sarcopenia: European consensus on definition and diagnosis: Report of the European Working Group on Sarcopenia in Older People. Age Ageing. 2010 Jul;39(4):412-23. doi: 10.1093/ageing/afq034. Epub 2010 Apr 13. PMID 20392703
- [Background] Rosenberg IH. Sarcopenia: origins and clinical relevance. J Nutr. 1997 May;127(5 Suppl):990S-991S. doi: 10.1093/jn/127.5.990S. PMID 9164280
- [Background] Baumgartner RN, Waters DL, Gallagher D, Morley JE, Garry PJ. Predictors of skeletal muscle mass in elderly men and women. Mech Ageing Dev. 1999 Mar 1;107(2):123-36. doi: 10.1016/s0047-6374(98)00130-4. PMID 10220041
- [Background] Janssen I, Heymsfield SB, Ross R. Low relative skeletal muscle mass (sarcopenia) in older persons is associated with functional impairment and physical disability. J Am Geriatr Soc. 2002 May;50(5):889-96. doi: 10.1046/j.1532-5415.2002.50216.x. PMID 12028177
- [Background] Goodpaster BH, Park SW, Harris TB, Kritchevsky SB, Nevitt M, Schwartz AV, Simonsick EM, Tylavsky FA, Visser M, Newman AB. The loss of skeletal muscle strength, mass, and quality in older adults: the health, aging and body composition study. J Gerontol A Biol Sci Med Sci. 2006 Oct;61(10):1059-64. doi: 10.1093/gerona/61.10.1059. PMID 17077199
- [Background] Roubenoff R. Sarcopenia and its implications for the elderly. Eur J Clin Nutr. 2000 Jun;54 Suppl 3:S40-7. doi: 10.1038/sj.ejcn.1601024. PMID 11041074
- [Background] Evans WJ, Campbell WW. Sarcopenia and age-related changes in body composition and functional capacity. J Nutr. 1993 Feb;123(2 Suppl):465-8. doi: 10.1093/jn/123.suppl_2.465. PMID 8429405
- [Background] Visser M, Pahor M, Taaffe DR, Goodpaster BH, Simonsick EM, Newman AB, Nevitt M, Harris TB. Relationship of interleukin-6 and tumor necrosis factor-alpha with muscle mass and muscle strength in elderly men and women: the Health ABC Study. J Gerontol A Biol Sci Med Sci. 2002 May;57(5):M326-32. doi: 10.1093/gerona/57.5.m326. PMID 11983728
- [Background] Peake J, Della Gatta P, Cameron-Smith D. Aging and its effects on inflammation in skeletal muscle at rest and following exercise-induced muscle injury. Am J Physiol Regul Integr Comp Physiol. 2010 Jun;298(6):R1485-95. doi: 10.1152/ajpregu.00467.2009. Epub 2010 Apr 14. PMID 20393160
- [Background] Paddon-Jones D, Sheffield-Moore M, Urban RJ, Sanford AP, Aarsland A, Wolfe RR, Ferrando AA. Essential amino acid and carbohydrate supplementation ameliorates muscle protein loss in humans during 28 days bedrest. J Clin Endocrinol Metab. 2004 Sep;89(9):4351-8. doi: 10.1210/jc.2003-032159. PMID 15356032
- [Background] Paddon-Jones D, Sheffield-Moore M, Aarsland A, Wolfe RR, Ferrando AA. Exogenous amino acids stimulate human muscle anabolism without interfering with the response to mixed meal ingestion. Am J Physiol Endocrinol Metab. 2005 Apr;288(4):E761-7. doi: 10.1152/ajpendo.00291.2004. Epub 2004 Nov 30. PMID 15572657
- [Background] Jensen GL. Inflammation: roles in aging and sarcopenia. JPEN J Parenter Enteral Nutr. 2008 Nov-Dec;32(6):656-9. doi: 10.1177/0148607108324585. PMID 18974248
- [Background] Evans WJ, Morley JE, Argiles J, Bales C, Baracos V, Guttridge D, Jatoi A, Kalantar-Zadeh K, Lochs H, Mantovani G, Marks D, Mitch WE, Muscaritoli M, Najand A, Ponikowski P, Rossi Fanelli F, Schambelan M, Schols A, Schuster M, Thomas D, Wolfe R, Anker SD. Cachexia: a new definition. Clin Nutr. 2008 Dec;27(6):793-9. doi: 10.1016/j.clnu.2008.06.013. Epub 2008 Aug 21. PMID 18718696
- [Background] Baumgartner RN, Koehler KM, Gallagher D, Romero L, Heymsfield SB, Ross RR, Garry PJ, Lindeman RD. Epidemiology of sarcopenia among the elderly in New Mexico. Am J Epidemiol. 1998 Apr 15;147(8):755-63. doi: 10.1093/oxfordjournals.aje.a009520. PMID 9554417
- [Background] Janssen I, Baumgartner RN, Ross R, Rosenberg IH, Roubenoff R. Skeletal muscle cutpoints associated with elevated physical disability risk in older men and women. Am J Epidemiol. 2004 Feb 15;159(4):413-21. doi: 10.1093/aje/kwh058. PMID 14769646
- [Background] Chumlea WC, Guo SS, Vellas B, Guigoz Y. Techniques of assessing muscle mass and function (sarcopenia) for epidemiological studies of the elderly. J Gerontol A Biol Sci Med Sci. 1995 Nov;50 Spec No:45-51. doi: 10.1093/gerona/50a.special_issue.45. PMID 7493217
- [Background] Paddon-Jones D, Short KR, Campbell WW, Volpi E, Wolfe RR. Role of dietary protein in the sarcopenia of aging. Am J Clin Nutr. 2008 May;87(5):1562S-1566S. doi: 10.1093/ajcn/87.5.1562S. PMID 18469288
- [Background] Volkert D, Berner YN, Berry E, Cederholm T, Coti Bertrand P, Milne A, Palmblad J, Schneider S, Sobotka L, Stanga Z; DGEM (German Society for Nutritional Medicine); Lenzen-Grossimlinghaus R, Krys U, Pirlich M, Herbst B, Schutz T, Schroer W, Weinrebe W, Ockenga J, Lochs H; ESPEN (European Society for Parenteral and Enteral Nutrition). ESPEN Guidelines on Enteral Nutrition: Geriatrics. Clin Nutr. 2006 Apr;25(2):330-60. doi: 10.1016/j.clnu.2006.01.012. PMID 16735082
- [Background] Milne AC, Potter J, Vivanti A, Avenell A. Protein and energy supplementation in elderly people at risk from malnutrition. Cochrane Database Syst Rev. 2009 Apr 15;2009(2):CD003288. doi: 10.1002/14651858.CD003288.pub3. PMID 19370584
- [Background] Flakoll P, Sharp R, Baier S, Levenhagen D, Carr C, Nissen S. Effect of beta-hydroxy-beta-methylbutyrate, arginine, and lysine supplementation on strength, functionality, body composition, and protein metabolism in elderly women. Nutrition. 2004 May;20(5):445-51. doi: 10.1016/j.nut.2004.01.009. PMID 15105032
- [Background] Malafarina V, Uriz-Otano F, Gil-Guerrero L, Iniesta R, Zulet MA, Martinez JA. Study protocol: High-protein nutritional intervention based on beta-hydroxy-beta-methylbutirate, vitamin D3 and calcium on obese and lean aged patients with hip fractures and sarcopenia. The HIPERPROT-GER study. Maturitas. 2013 Oct;76(2):123-8. doi: 10.1016/j.maturitas.2013.06.016. Epub 2013 Jul 26. PMID 23891440
- [Background] Malafarina V, Uriz-Otano F, Iniesta R, Gil-Guerrero L. Effectiveness of nutritional supplementation on muscle mass in treatment of sarcopenia in old age: a systematic review. J Am Med Dir Assoc. 2013 Jan;14(1):10-7. doi: 10.1016/j.jamda.2012.08.001. Epub 2012 Sep 13. PMID 22980996
- [Background] Malafarina V, Uriz-Otano F, Iniesta R, Gil-Guerrero L. Sarcopenia in the elderly: diagnosis, physiopathology and treatment. Maturitas. 2012 Feb;71(2):109-14. doi: 10.1016/j.maturitas.2011.11.012. Epub 2011 Dec 6. PMID 22153348
- [Derived] Malafarina V, Uriz-Otano F, Malafarina C, Martinez JA, Zulet MA. Effectiveness of nutritional supplementation on sarcopenia and recovery in hip fracture patients. A multi-centre randomized trial. Maturitas. 2017 Jul;101:42-50. doi: 10.1016/j.maturitas.2017.04.010. Epub 2017 Apr 22. PMID 28539168